CLINICAL TRIAL: NCT02299102
Title: A Study Comparing Powered Ported Bone Marrow Aspiration Procedures to Manual Standard Bone Marrow Aspiration Procedures Using Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vidacare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2014-12
Record Dates: First submitted 2014-11-17; First posted 2014-11-24 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: Aspiration Procedures; Bone Marrow; To compare powered ported bone marrow aspiration procedures to manual standard bone marrow aspiration procedures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Jamshidi Manual Standard Device (Other): The Jamshidi manual standard device will be randomized for use on the right or left iliac crest
  Interventions: Device: Jamshidi Manual Standard Device
- OnControl Powered Ported Device (Other): The OnControl power ported device will be used on the opposite iliac crest
  Interventions: Device: OnControl Powered Ported Device

INTERVENTIONS:
Device: Jamshidi Manual Standard Device — Jamshidi Manual Standard Device
  Arms: Jamshidi Manual Standard Device
Device: OnControl Powered Ported Device — OnControl Powered Ported Device
  Arms: OnControl Powered Ported Device

SUMMARY:
This single center, randomized, controlled trial will compare the manual standard bone marrow aspiration device to the powered ported bone marrow aspiration device for use in the iliac crest in healthy adult volunteers. The study will compare the subjects' perceived level of pain, time to sample acquisition, and quality of specimen yield of these devices. To serve as their own control, each subject will receive bilateral bone marrow aspiration procedures using both the manual standard and powered ported devices.

DETAILED DESCRIPTION:
This single center, randomized, controlled trial will compare the manual standard bone marrow aspiration needle to the power ported aspiration needle for use in the posterior iliac crest of healthy volunteers for bone marrow aspiration specimen collection. The study will compare the quality of specimen yield of the devices, subject reported level of pain with needle insertion and aspiration, and time from needle/skin contact to needle insertion and to sample acquisition. Each subject will serve as his/her own control and will receive bilateral bone marrow aspiration procedures using both the manual standard and power ported needles. The order in which the devices are used for each subject's procedures and on which side each device will be used will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Adults 21 years of age and over
* Able to lay flat in prone position on a table for up to 1 hour
* Self-reported as healthy, as confirmed by the investigator during the medical history review and physical examination
* Female subjects with a negative urine pregnancy test at screening visit

Exclusion Criteria:

* Reported fever within 7 days of the screening visit
* Reported active infection within 7 days of the screening visit
* Fever on day of study procedure
* Signs/symptoms of active infection on day of study procedure
* Imprisoned
* Self identified as pregnant or lactating
* Cognitively impaired
* Patients with one or more conditions precluding bone marrow aspiration
* Excessive tissue and/or absence of adequate anatomical landmarks in target bone
* Allergy to local anesthetics
* Unable to lay flat in prone position
* Prothrombin time and International Normalized Ratio (PT/INR) results outside of normal range on screening lab work and deemed clinically significant by the investigator

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Quality of aspirate specimen yield | 30 days
  Determined by a pathologist unaware of the device type used to obtain the specimen. The stained bone marrow aspirate smears will be evaluated for the presence of bone marrow particles (spicules) as well as the relative cellularity and quality of the bone marrow cells present in the smears.

SECONDARY OUTCOMES:
Subject reported level of pain with needle insertion | 1 Day
  The secondary objective of this study is to compare the procedure of bone marrow aspiration for procedure time and subject reported level of pain when performed using the power ported and the manual standard aspiration needles.
Subject reported level of pain with aspiration | 1 Day
  The secondary objective of this study is to compare the procedure of bone marrow aspiration for procedure time and subject reported level of pain when performed using the power ported and the manual standard aspiration needles.
Time from needle/periosteum contact to needle insertion through the cortex | 1 Day
  The secondary objective of this study is to compare the procedure of bone marrow aspiration for procedure time and subject reported level of pain when performed using the power ported and the manual standard aspiration needles.
Time from needle/periosteum contact to removal of the needle following sample acquisition | 1 Day
  The secondary objective of this study is to compare the procedure of bone marrow aspiration for procedure time and subject reported level of pain when performed using the power ported and the manual standard aspiration needles.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Therapy and Research LLC., San Antonio, Texas, United States